CLINICAL TRIAL: NCT07212452
Title: Tranexamic Acid : Nebulization vs IV Route for Hemoptysis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Laiba Qamar, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #NTranexamic#
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Hemoptysis; NEBULIZATION; Tranexamic Acid
Keywords: Hemoptysis; Nebulization; tranexamic acid
MeSH Terms: conditions — Hemoptysis | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: The intervention will be given to the participants via providing the tranexamic acide through both IV and nebulization routes.
Masking Description: There is no masking as the participnats will be explained the whole process and consent would be taken for using the either route for administration of tranexamic acid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group receiving tranexamic acid via IV route (Active Comparator): Tranexamic acid has been used conventionally for hemoptysis via IV route
  Interventions: Drug: Tranexamic Acid (TXA)
- The Group receiving tranexamic acid via nebulization (Experimental): Tranexamic acid when given through nebulization can be more effective than IV route in controlling hemoptysis
  Interventions: Drug: Tranexamic Acid (TXA)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — In this study we are comparing the effect of tranexamic acid on hemoptysis when given through IV route and nebulization
  Other Names: nebulization

SUMMARY:
This study compares the effect of tranexamic acid on hemoptysis when given through the conventional IV route and Through nebulization.

DETAILED DESCRIPTION:
The investigators are conducting a randomized controlled trial for the comparison of routes through which tranexamic acid can be given to control hemoptysis. The study participants will be divided into 2 groups randomly and 1 group will be assigned to use IV route while other will be assigned the nebulization route and the result variables include the time taken for complete control of hemoptysis and recurrence time. Another variable is the reduction in amout of blood in sputum after each intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mild to moderate hemoptysis < 600ml/ 24 hours of age 12 to 80 years and both genders.
2. Patients with hemoptysis due to infective pathology.
3. Patients with hemoptysis due to malignant pathology.

Exclusion Criteria:

1. Patients on antiplatelet therapy or aspirin
2. Hemoptysis after penetrating lung injury e.g. firearm injury
3. Patients with history of asthma

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Time to control hemoptysis | 48 hours
  In this study the time taken by tranexamic acid to acehive comolete control of hemoptysis will be compared when given through IV and nebulization.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gopinath B, Mishra PR, Aggarwal P, Nayaka R, Naik SR, Kappagantu V, Shrimal P, Ramaswami A, Bhoi S, Jamshed N, Sinha TP, Ekka M, Kumar A. Nebulized vs IV Tranexamic Acid for Hemoptysis: A Pilot Randomized Controlled Trial. Chest. 2023 May;163(5):1176-1184. doi: 10.1016/j.chest.2022.11.021. Epub 2022 Nov 19. PMID 36410494
- See also: The sample article is available through this link — https://pubmed.ncbi.nlm.nih.gov/36410494/